CLINICAL TRIAL: NCT03869723
Title: Evaluation of Virtual Surgical Planning Systems and Customized Devices in Fibula Free Flap Mandibular Recontruction
Brief Title: Virtual Surgical Planning Systems in Mandibular Reconstruction
Acronym: VP3D
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2019_002
Record Dates: First submitted 2019-02-08; First posted 2019-03-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Mandibular Neoplasms
MeSH Terms: conditions — Mandibular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional surgery: Classical surgery for mandibular reconstruction with fibula free flap
  Interventions: Procedure: Conventional surgery
- Virtual planning: Fibula free flap in mandibular reconstruction using preoperative virtual planning, cutting guides and osteosynthesis plates. Preoperative modeling was conducted by obtaining scans of patient maxillofacial skeleton and angioscans of the lower extremities. The planning phase was then carried out by the surgeon and the engineer (from MATERIALISE, Leuven, Belgium) so as to define the clinical and technical parameters of the reconstruction. This stage consisted of discussing and determining osteotomy lines, donor side, anastomosis site, and overall reconstruction contour. Resection was decided by the surgeon. 3D modeling and the manufacture of cutting guides and customized osteosynthesis plates were then undertaken
  Interventions: Procedure: Virtual planning using customized surgical devices

INTERVENTIONS:
Procedure: Virtual planning using customized surgical devices — Preoperative modeling was conducted by obtaining scans of patient maxillofacial skeleton and angioscans of the lower extremities. The planning phase was then carried out by the surgeon and the engineer (from MATERIALISE, Leuven, Belgium) so as to define the clinical and technical parameters of the reconstruction. This stage consisted of discussing and determining osteotomy lines, donor side, anastomosis site, and overall reconstruction contour. Resection was decided by the surgeon. 3D modeling and the manufacture of cutting guides and customized osteosynthesis plates were then undertaken
  Groups: Virtual planning
Procedure: Conventional surgery — Classical surgery for mandibular reconstruction with fibula free flap
  Groups: Conventional surgery

SUMMARY:
The purpose of this study was to evaluate the accuracy of virtual planning using customized surgical devices (VP3D) in fibula free flap mandibular reconstruction. Virtual planning was compared to postoperative scans using cephalometric and three-dimensional (3D) measurements. Operative times of both VP3D and conventional surgery groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent fibula free flap for mandibular reconstruction
* Patient ≥18 years old
* patient alive 6 months after completion of treatment

Exclusion Criteria:

* Patient without post-operative scan evaluation
* Patient with a chirurgical contraindication
* Pregnant or nursing woman
* Adult requiring protection (guardianship, supervision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent fibula free flap for mandibular reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the cephalometrics measurements between the virtual model and postoperative outcomes | Six months after surgery
  The virtual model obtained using preoperative surgical planning will be compared with postoperative outcomes derived from facial bone scans conducted on all VP3D group patients 6 months after surgery (MIMICS INNOVATION suite 2.1 software, MATERIALISE, Leuven, Belgium).
  The cephalometrics measurements (in mm) between the virtual model and postoperative outcomes will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanc J, Fuchsmann C, Nistiriuc-Muntean V, Jacquenot P, Philouze P, Ceruse P. Evaluation of virtual surgical planning systems and customized devices in fibula free flap mandibular reconstruction. Eur Arch Otorhinolaryngol. 2019 Dec;276(12):3477-3486. doi: 10.1007/s00405-019-05625-z. Epub 2019 Sep 9. PMID 31501989